CLINICAL TRIAL: NCT02078063
Title: Mepivacaine for Pain Relief at Insertion of Intrauterine Contraception
Brief Title: Analgesia for Insertion of Intrauterine Contraception
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Helena Kopp Kallner, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WIUC13 version II
Record Dates: First submitted 2013-11-21; First posted 2014-03-05 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Insertion of Intrauterine Contraception
MeSH Terms: interventions — Mepivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepivacaine (Experimental): 10 ml of Mepivacaine for injection (Carbocain®) 10 mg/ml instilled into the uterus through a hydrosonography catheter
  Interventions: Drug: Mepivacaine
- NaCL (Placebo Comparator): 10 ml NaCl 9mg/ml instilled into the uterus through a hydrosonography catheter
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mepivacaine — 10 ml of Mepivacaine for injection (Carbocain®) 10 mg/ml instilled into the uterus through a hydrosonography catheter
  Other Names: Carbocain (R)
  Arms: Mepivacaine
Drug: Placebo — 10 ml of NaCl 0.9 mg/ml instilled into the uterus through a hydrosonography catheter
  Arms: NaCL

SUMMARY:
Use of long acting reversible contraception (LARC) such as implants or intrauterine contraception (IUC) has been shown to reduce repeat abortions. LARCs have the advantage of being independent of user error and are considered to be underused, especially among young individuals where oral methods have high rates of user failure. IUC is often underused in young or nulliparous women due to fear of pain at insertion.

10 ml of mepivacaine (10mg/ml) or 10ml of sodium hydrochloride will be injected into the uterine cavity through a hydrosonography catheter before the tenaculum has been applied but prior to sounding and to insertion of the IUC.

The investigators' hypothesis is that instillation of 10 ml (10mg/ml) mepivacaine though a hydrosonography catheter prior to any instrument placement will provide more effective pain relief than instillation of 10 ml placebo (sodium chloride 9mg/ml).

Primary objective: To evaluate the difference in pain score at the time of the insertion of the IUC between treatment and control group.

Secondary objectives: To evaluate acceptability of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age and
* opting for IUC for contraception
* with a negative pregnancy test
* willing to participate in the study after it has been explained orally and in written

Exclusion Criteria:

* previous conisation,
* known cervical stenosis,
* signs of ongoing genital infection,
* known uterine abnormality,
* any condition resulting in bleeding disorder or contraindication to any local anestetic will be excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-11; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
pain | On day of insertion
  difference in pain score (VAS)at the time of the insertion of the IUC between treatment and control group.

SECONDARY OUTCOMES:
Acceptability | 30 minutes after insertion
  They will be asked if the would opt to have this type of pain relief were the ever to insert a new IUC (yes/no), if they would recommend this type of pain relief to any other women (yes/no) and to state how the procedure was compared to their expectations (worse/as expected/better).

CONTACTS AND LOCATIONS:
Overall Officials: Helena Kopp Kallner, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - Dept of Obstetrics and Gynecology, Danderyd Hospital, Stockholm
  - Upplands Väsby Ungdomsmottagning, Stockholm

REFERENCES:
- [Derived] Envall N, Lagercrantz HG, Sunesson J, Kopp Kallner H. Intrauterine mepivacaine instillation for pain relief during intrauterine device insertion in nulliparous women: a double-blind, randomized, controlled trial. Contraception. 2019 Jun;99(6):335-339. doi: 10.1016/j.contraception.2019.02.003. Epub 2019 Mar 1. PMID 30831101